CLINICAL TRIAL: NCT06888908
Title: Perioperative Change in Blood Volume and Fluid Distribution in Total Hip Arthroplasty
Brief Title: Changes in Perioperative Blood Volume and Fluid Distribution in Patients Undergoing Primary Total Hip Replacement.
Status: Recruiting | Type: Observational
Sponsor: Copenhagen University Hospital, Hvidovre (Other)
Responsible Party: Principal Investigator, Puk Kristiansen, MD, Ph.d.-student, Copenhagen University Hospital, Hvidovre
Other Study IDs: H-24062107
Record Dates: First submitted 2025-03-08; First posted 2025-03-21 (Actual); Last update posted 2025-03-21 (Actual); Status verified 2025-03

CONDITIONS: Hip Arthroplasty Replacement
Keywords: Blood loss; Blood volume
MeSH Terms: conditions — Hemorrhage

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
Clinical assessment of bleeding and calculation of perioperative blood loss do not provide an accurate estimate of blood volume. This makes rational fluid management difficult, which is of high importance for patient-related outcomes. The availability of carbon monoxide(CO)-rebreathing allows for simple, non-invasive and precise measurement of changes in blood volume.

The purpose of the study is to investigate and describe changes in blood volume and fluid distribution perioperative in patients undergoing total hip arthroplasty. Furthermore, to investigate the association between changes in blood volume and incidence of orthostatic insufficiency.

ELIGIBILITY:
Inclusion Criteria:

* Patients scheduled for an elective total hip arthoplasty (THA) in a standardized fast track setting.
* Capable of participating in CO-rebreathing measurement
* Age ≥ 18 years
* Able to speak and understand Danish
* Has provided written informed consent.

Exclusion Criteria:

* Intraoperative blood loss exceeding 750 mL.
* Perioperative need for a blood transfusion.
* Confirmed or suspected coagulopathies.
* Factors that make CO-rebreathing measurement impossible.
* Known orthostatic intolerance.
* American Society of Anesthesiologists physical status (ASA) classification ≥ 4.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients scheduled for an elective total hip arthoplasty (THA) at Hvidovre University Hospital and undergo the proceduce under spinal anesthesia with propofol sedation.
Sampling Method: Probability Sample
Enrollment: 25 (Estimated)
Dates: Start 2025-03 (Estimated); Primary Completion 2026-09 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Change in total blood volume (TBV) | Preoperatively and 6 hours postoperatively
  Measured in milliliter (mL)

SECONDARY OUTCOMES:
Change in total blood volume (TBV) | Preoperatively and 24 hours postoperatively
  measured in mL
Changes in total hemoglobin mass (tHgb) | Preoperatively, 6 hours postoperatively and 24 hours postoperatively
  Measured in gram (g)
Changes in erythrocyte volume (EBV) | Preoperatively, 6 hours postoperatively and 24 hours postoperatively
  Measured in mL
Changes in plasma volume (PV) | Preoperatively, 6 hours postoperatively and 24 hours postoperatively
  Measured in mL
Changes in hematokrit (Ht) | Preoperatively, 6 hours postoperatively and 24 hours postoperatively
  Reported as percentage(%)
Changes in hemoglobin (Hg) concentration | Preoperatively, 6 hours postoperatively and 24 hours postoperatively
  Measured in millimoles/liter(mmol/L)
Changes in Total body water(TBW), intra-(ICF) and extracellular(ECF) fluid distribution | Preoperatively, 6 hours postoperatively and 24 hours postoperatively
  Full body water via bioelectrical impedance analysis. The individual components are reported in L and percent.
Changes in C-Reactive Protein (CRP) | Preoperatively, 6 hours postoperatively and 24 hours postoperatively
  Measured in milligram/liter (mg/L)
Incidence of orthostatic intolerance during mobilization | Preoperatively, 6 hours postoperatively and 24 hours postoperatively
  Symptoms of orthostatic intolerance: dizziness, nausea, vomiting, blurry vision or syncope during mobilization
Association between total blood loss and incidence of orthostatic intolerance | Preoperatively, 6 hours postoperatively and 24 hours postoperatively
  Blood loss measured in mL. Symptoms of orthostatic intolerance: dizziness, nausea, vomiting, blurry vision or syncope during mobilization
Association between changes in C-Reactive Protein and total blood loss | Preoperatively, 6 hours postoperatively and 24 hours postoperatively
  C-Reactive Protein measured in mg/L and total blood loss measured in mL
Association between peripheral perfusion index and total blood loss | Preoperatively, 6 hours postoperatively and 24 hours postoperatively
  Peripheral perfusion index measured in percent and total blood loss in mL
Association between total hemoglobin (SpHb) and total blood loss | Preoperatively, 6 hours postoperatively and 24 hours postoperatively
  SpHb measured as gram/deciliter and total blood loss measured in mL

OTHER OUTCOMES:
Intraoperativ estimation of bleeding | Intraoperative at end of the surgical procedure
  Measured by weighting gauze (gram)
Intraoperative bleeding | Intraoperative at end of the surgical procedure
  Measured by visual estimation in surgical drains (mL)

CONTACTS AND LOCATIONS:
Overall Officials: Nicolai Foss, Professor, Dr. Med., Study Director — Department of Anesthesiology and Intensive Care Medicine, Copenhagen University Hospital, Hvidovre
Locations (1):
- Hvidovre University Hospital, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: No